CLINICAL TRIAL: NCT03731468
Title: Effect of Dexmethasone Addition to Bupivacaine in Bilateral Intermediate Cervical Block in Thyroid Surgery
Brief Title: Ultrasound Guided Intermediate Cervical Plexus Block in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UDLC
Record Dates: First submitted 2018-07-09; First posted 2018-11-06 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, Local; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmethasone group (Active Comparator): 8 mg dexamethasone will be added to local anaesthetics
  Interventions: Drug: Dexamethasone
- control group (Sham Comparator): isobaric bupivacaine will be given on each side
  Interventions: Drug: local anesthetic

INTERVENTIONS:
Drug: local anesthetic — ultrasound guided superficial cervical block in thyroid surgery
  Arms: control group
Drug: Dexamethasone — dexamethasone will be added to ultrasound guided superficial cervical block in thyroid surgery
  Arms: dexmethasone group

SUMMARY:
studying the effect of dexmeditomidine addition to bupivacaine in bilateral intermediate cervical block for patients undergoing thyroidectomy under general anaesthesia

DETAILED DESCRIPTION:
80 patients who will be undergoing elective thyroidectomy will be randomly allocated into one of two groups ; group A will receive 20 mg isobaric bupivacaine + 8 mg dexamethasone(diluted in 5 ml) group B will receive 20 mg isobaric bupivacaine + 1 ml normal saline. block will be done under complete a septic condition after induction of general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* ASA 1, II, AND III

Exclusion Criteria:

* Patient refusal
* Infection at the entry site
* BMI > 3

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia duration | 24 hour postoperative
  time of first analgesic requirement is the time of end of block analgesia

SECONDARY OUTCOMES:
postoperative complications related to the block | 8 hours
  occurrence of complications secondary to the block well be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt